CLINICAL TRIAL: NCT00789867
Title: Evaluation of Safety and Gene Expression With a Single Dose of pGM169/GL67A Administered to the Nose and Lung of Individuals With Cystic Fibrosis
Brief Title: Single Dose of pGM169/GL67A in CF Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); University of Oxford (Other); University of Edinburgh (Other); Cystic Fibrosis Trust (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cro851
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cystic Fibrosis
Keywords: Single dose; Pilot; Safety; Gene expression; Tolerability; CFTR gene; Cystic fibrosis; Non-viral
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20ml pGM169/GL67A (Experimental): Received a nebulized dose 20ml via an breath-actuated nebulizer
  Interventions: Drug: pGM169/GL67A
- 10ml pGM169/GL67A (Experimental): Received a nebulized dose 10ml via an breath-actuated nebulizer
  Interventions: Drug: pGM169/GL67A
- 5ml pGM169/GL67A (Experimental): Received a nebulized dose 5ml via an breath-actuated nebulizer
  Interventions: Drug: pGM169/GL67A

INTERVENTIONS:
Drug: pGM169/GL67A — Received a nebulized dose via an breath-actuated nebulizer
  Other Names: 5ml pGM169/GL67A, 10ml pGM169/GL67A and 20ml pGM169/GL67A

SUMMARY:
The study objectives are to assess safety, tolerability and gene expression after a single dose of non-viral CFTR gene therapy (pGM169/GL67A) administered to the nose and lungs of patients with cystic fibrosis.

DETAILED DESCRIPTION:
The trial is designed as single administration to nose and lung. Initially, in Part A, 3 patients will be dosed individually one week apart with 10 ml (26.5mg pDNA) via nebuliser and a nasal dose equivalent to 10% of this (based on relative surface area calculations: conducting airways approximate 540 cm2; nasal epithelium from both nostrils approximately 40 cm2). Based on our previous study, we do not expect any side effects of the nasal dose, but we are taking this opportunity, as this group will not be undergoing bronchoscopic efficacy measures, to assess gene transfer to the nasal epithelium. A further group of 3 patients will then be treated in exactly the same way with 20 ml nebulised and a 2 ml nasal dose.

Subsequently, patients will receive doses of 2 ml (nasal) and 20 ml (nebulised). These patients will undergo more intensive monitoring for gene expression both before and after administration.

In Part B of the protocol, we will test combinations of delivery conditions and dose in an attempt to identify the maximal tolerated dose. We may also use Ibuprofen or Prednisolone in standard clinical doses around the dosing period to reduce the inflammatory response. Delivery conditions include: standard nebulisation (each 5 ml over 25 minutes as in Part A), slow (each 5 ml over 75-150 minutes) and divided (standard rate delivery with a period of up to 6 hours between aliquots). With these conditions we will test the following doses until a tolerable dose is reached: 20 ml (no standard delivery as sufficient data already available from Part A); 10 ml; 5 ml; 2.5 ml. Each dosing strategy will initially be performed in a cohort of 3 patients although numbers may need to be increased to 6 if data are inconclusive. Once a satisfactory Single dose of pGM169/GL67A in CF patients; cro851 Version 10; 16.08.2010 10 dose and nebulisation strategy has been identified, the numbers receiving this will be increased to 6. The maximum number of patients recruited to this arm of the study will be 30. Part B will also allow either these subjects or others to receive a 2 ml nasal dose with both pre and post-measurements of nasal PD.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis confirmed by sweat testing or genetic analysis
* Males and females aged 16 years and above
* Forced expiratory volume in the 1st second (FEV1) > 60% predicted values
* Clinical stability at entry
* Prepared to take effective contraceptive precautions for the duration of their participation in the study and for 3 months thereafter
* If taking regular rhDNase (pulmozyme) is willing, and considered able by independent medical carers, to withhold treatment for 24 hours before and 24 hours after the gene therapy dose
* Written informed consent obtained
* Permission to inform GP of participation in study

Exclusion Criteria:

* Infection with Burkholderia cepacia complex organisms or MRSA
* Significant nasal pathology including polyps, clinically-significant rhinosinusitis, or recurrent severe epistaxis (nose bleeds)
* Acute upper respiratory tract infection within the last 2 weeks
* Previous spontaneous pneumothorax without pleurodesis
* Recurrent severe haemoptysis
* Current smoker
* Significant comorbidity including:

  1. Moderate/severe CF liver disease
  2. Significant renal impairment
  3. Significant coagulopathy
* Receiving 2nd line immunosuppressant drugs such as methotrexate, cyclosporine, intravenous immunoglobulin preparations
* Pregnant or breastfeeding

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Alton, Study Director — Imperial College London; Jane C Davies, Principal Investigator — Imperial College London; Uta Griesenbach, Principal Investigator — Imperial College London; Steve Hyde, Principal Investigator — University of Oxford; Deborah Gill, Principal Investigator — University of Oxford; David Porteous, Principal Investigator — Edinburgh University; Chris Boyd, Principal Investigator — Edinburgh University; Alastair Innes, Principal Investigator — Edinburgh University
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alton EW, Stern M, Farley R, Jaffe A, Chadwick SL, Phillips J, Davies J, Smith SN, Browning J, Davies MG, Hodson ME, Durham SR, Li D, Jeffery PK, Scallan M, Balfour R, Eastman SJ, Cheng SH, Smith AE, Meeker D, Geddes DM. Cationic lipid-mediated CFTR gene transfer to the lungs and nose of patients with cystic fibrosis: a double-blind placebo-controlled trial. Lancet. 1999 Mar 20;353(9157):947-54. doi: 10.1016/s0140-6736(98)06532-5. PMID 10459902
- [Result] Alton EW, Boyd AC, Porteous DJ, Davies G, Davies JC, Griesenbach U, Higgins TE, Gill DR, Hyde SC, Innes JA; UK Cystic Fibrosis Gene Therapy Consortium *. A Phase I/IIa Safety and Efficacy Study of Nebulized Liposome-mediated Gene Therapy for Cystic Fibrosis Supports a Multidose Trial. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1389-92. doi: 10.1164/rccm.201506-1193LE. No abstract available. PMID 26623687
- See also: UK CF Gene Therapy Consortium website — http://www.cfgenetherapy.org.uk/

RESULTS

PARTICIPANT FLOW:
Groups:
- 20 ml pGM169/GL67A: Received a nebulized dose 20ml via an breath-actuated nebulizer
Period: Overall Study
Arm/Group | 20 ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
Started | 17 | 10 | 8
Completed | 17 | 10 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A | Total
Number analyzed (Participants) | 17 | 10 | 8 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 2
  Between 18 and 65 years | 16 | 9 | 8 | 33
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 26.7 [17.3 to 50.1] | 33.2 [16.4 to 61.6] | 32.6 [24.3 to 46.4] | 27.4 [16.4 to 61.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 12
  Male | 12 | 6 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United Kingdom | 17 | 10 | 8 | 35

OUTCOME MEASURES:

1. Primary Outcome: Body Maximum Temperature
Time Frame: 6-8h
Population: A lower number of participants due to missing data
Measure: Mean (Standard Deviation); unit: celsius
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
Number analyzed (Participants) | 15 | 6 | 6
celsius | 38.6 (0.5) | 38.0 (0.7) | 37.4 (0.3)
Statistical Analysis 1: Comparison: 20ml pGM169/GL67A vs 10ml pGM169/GL67A vs 5ml pGM169/GL67A; Test type: Other; p = 0.0002, Kruskal-Wallis

2. Primary Outcome: Blood Leukocytes
Description: Blood leukocytes measure
Time Frame: 8h
Population: A lower number of participants due to missing data
Measure: Mean (Standard Deviation); unit: x1000000000 cells/L
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
Number analyzed (Participants) | 15 | 6 | 6
x1000000000 cells/L | 15.8 (3.2) | 14.1 (4.5) | 12.8 (3.8)
Statistical Analysis 1: Comparison: 20ml pGM169/GL67A vs 10ml pGM169/GL67A vs 5ml pGM169/GL67A; Test type: Other; p = 0.22, Kruskal-Wallis

3. Primary Outcome: Blood Neutrophils
Description: Blood neutrophils measures
Time Frame: 8h
Population: A lower number of participants due to missing data
Measure: Mean (Standard Deviation); unit: 1000000000/L
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
Number analyzed (Participants) | 15 | 6 | 6
1000000000/L | 13.9 (3.4) | 11.3 (4.1) | 9.8 (3.5)
Statistical Analysis 1: Comparison: 20ml pGM169/GL67A vs 10ml pGM169/GL67A vs 5ml pGM169/GL67A; Test type: Other; p = 0.06, Kruskal-Wallis

4. Primary Outcome: FEV1 Relative % Drop
Description: FEV1 relative % drop measure
Time Frame: 8h
Population: A lower number of participants due to missing data
Measure: Mean (Standard Deviation); unit: % of drop
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
Number analyzed (Participants) | 15 | 6 | 6
% of drop | 24.6 (9.3) | 17.5 (7.8) | 16.8 (4.0)
Statistical Analysis 1: Comparison: 20ml pGM169/GL67A vs 10ml pGM169/GL67A vs 5ml pGM169/GL67A; Test type: Other; p = 0.08, Kruskal-Wallis

5. Primary Outcome: FVC Relative % Drop
Description: FVC relative % drop measure
Time Frame: 6h
Population: A lower number of participants due to missing data
Measure: Mean (Standard Deviation); unit: % drop
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
Number analyzed (Participants) | 15 | 6 | 6
% drop | 20.7 (2.9) | 13.7 (2.2) | 14.7 (2.2)
Statistical Analysis 1: Comparison: 20ml pGM169/GL67A vs 10ml pGM169/GL67A vs 5ml pGM169/GL67A; Test type: Other; p = 0.22, Kruskal-Wallis

6. Primary Outcome: Lung Clearance Index - LCI
Description: Lung clearance index measure is a measure of abnormal ventilation distribution derived from the multiple breath inert gas washout technique.
Time Frame: 8h
Population: A lower number of participants due to missing data
Measure: Mean (Standard Deviation); unit: index
Groups:
- 20ml pGM169/GL67A: Received a nebulized dose 20ml via an breath-actuated nebulizer nebulizer
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
Number analyzed (Participants) | 15 | 6 | 6
index | 0.75 (0.3) | 0.32 (0.1) | 0.32 (.01)
Statistical Analysis 1: Comparison: 20ml pGM169/GL67A vs 10ml pGM169/GL67A vs 5ml pGM169/GL67A; Test type: Other; p = 0.003, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | 20ml pGM169/GL67A | 10ml pGM169/GL67A | 5ml pGM169/GL67A
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 14/17 | 7/10 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20ml pGM169/GL67A (N=17) | 10ml pGM169/GL67A (N=10) | 5ml pGM169/GL67A (N=8)
Acute pancreatitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Injury in luvula sustained from pressure of tube during bronchoscopy 03/04/2009 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20ml pGM169/GL67A (N=17) | 10ml pGM169/GL67A (N=10) | 5ml pGM169/GL67A (N=8)
Mild self limiting influenza like systemic response (Immune system disorders) | 14 (14) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes